CLINICAL TRIAL: NCT04238728
Title: An Unblinded, Open-label Study Evaluating the Safety of Silverlon to Manage Radiation Dermatitis.
Brief Title: Silverlon to Reduce Radiation Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julie Ryan Wolf, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00004587
Record Dates: First submitted 2020-01-16; First posted 2020-01-23 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Intervention Model Description: Silverlon dressing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Silverlon arm (Experimental): Silverlon is a silver-nylon dressing approved for treatment of burns and wounds. In this study, the Silverlon dressing will be applied to the whole breast area receiving radiation therapy throughout the prescribed course of radiation therapy starting the first day of radiation therapy and until two weeks post-radiation. The Silverlon dressing will be held in place by a bra and worn daily except when bathing/showering, received radiation therapy, or swimming. Subject document when they remove the dressing and apply the dressing every day.
  Interventions: Device: Silverlon

INTERVENTIONS:
Device: Silverlon — silver nylon dressing will be applied daily

SUMMARY:
The purpose of this study is to see if a silver-nylon dressing (Silverlon®, Argentum Medical) is useful for the prevention or treatment of radiation dermatitis in patients receiving radiation therapy to the breast.

ELIGIBILITY:
Inclusion Criteria:

* Females, 22 years of age or older, with diagnosis of primary breast cancer (excluding inflammatory and medullary breast cancers).
* Scheduled to receive short-course external beam radiation therapy (i.e., 2.0-3.0 Gy for 15-20 fractions) or conventional external beam radiation therapy (i.e., 1.8-2.0 Gy for 25-40 fractions), with or without boost dose, to the whole breast.
* Not receiving concurrent chemotherapy.
* Subject may have had chemotherapy prior to radiation. A minimum of two weeks is required between the end of chemotherapy and start of radiation therapy.
* No history of previous breast or chest radiation therapy.
* Subject may or may not have had surgery (lumpectomy or mastectomy) prior to RT. (Note: Surgery is not required for eligibility).
* Subjects may be currently prescribed hormone treatment or Herceptin therapy.
* Subjects must be able to read, speak, and understand English language (all study forms are in English).
* Subjects must be able to give informed consent.
* Subjects must be willing to have photographs taken of radiation-induced skin changes in the radiation treatment area.
* Subjects must be willing to wear Silverlon dressing and undergarment (i.e., bra) at all times, except when bathing/showering and during their radiation therapy session.
* Subjects must be willing to complete a Silverlon Compliance Log to document the date and time that Silverlon was removed and applied each day during the study.

Exclusion Criteria:

* Diagnosis of medullary or inflammatory breast cancer.
* Diagnosis of tumors of the breast other than primary breast cancer (skin cancers, lymphomas, or metastatic cancers from other primary sites).
* Partial breast irradiation (PBI) treatment technique is not eligible.
* Concurrent chemotherapy.
* Pregnant or planning to become pregnant. Pregnant females are ineligible because pregnancy is a contraindication for RT. All subjects of childbearing potential will be asked if they are pregnant or could be pregnant. The subject must respond "no" to continue with radiation and to participate in this clinical study.
* Previous radiation to the chest or breast.
* Radiation being given for palliative purposes.
* Presence of unhealed surgical wounds, biopsy sites, open wounds in the breast or chest area.
* Presence of breast infection.
* Subjects currently on anti-EGFR (human epidermal growth factor receptor) therapy, such as Iressa (gefitinib) or Erbitux (cetuximab, C225).
* Previous diagnosis of autoimmune disease, connective tissue disease, or radiosensitivity disorder.
* Presence of any active dermatological issues in radiation treatment area (i.e., fungal skin infection, dermatitis, psoriasis plaques, etc).
* Chronic skin disease of the breast, previous breast trauma or scarring of the breast
* Subjects with known sensitivity to silver or nylon.
* Subjects unable or unwilling to wear Silverlon dressings and undergarment (i.e., bra) at all times, except while bathing/showering and during their radiation therapy session.
* Subjects unable to speak, read, or understand English language (all study forms are in English).

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subjects must be female. Approximately 99% of breast cancer diagnoses occur in adult women. Since too few men are diagnosed with the disease to allow meaningful sub-group analyses, subject accrual will only be women (≥ 18 years of age) with breast cancer. Additionally, men are unlikely to wear a bra and the dressing would have to be held in place using another method, which is not the purpose of this study.
Enrollment: 31 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wilmot Cancer Institute, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be shared if requested.
Supporting Information: Study Protocol, SAP, ICF

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 111 patient screened. 41 were ineligible. 31 were not approached because they already started radiation therapy or were undergoing chemotherapy or surgery. 39 were approached. 1 screen failed and 31 consented and started the intervention.
Period: Overall Study
Arm/Group | Silverlon Arm
Started | 31
Completed | 28
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Silverlon Arm
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Skin Event
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Silverlon Arm
Number analyzed (Participants) | 28
Participants | 1

2. Secondary Outcome: Number of Participants With Each Grade of the Radiation Therapy Oncology Group (RTOG) Toxicity Score
Description: The radiation oncologist or nurse will rate the skin reaction in the area where Silverlon dressing was applied using the RTOG scale which ranges from 0-5 with higher scores indicating worse outcome.
  Grade 0 No change; Normal Skin Grade 1 Faint erythema; dry desquamation; epilation, decreased sweating Grade 2 Tender or bright erythema; moderate edema; patchy moist desquamation only in skin folds.
  Grade 3 Confluent moist desquamation in areas other than skin folds; pitting edema Grade 4 Ulceration; hemorrhage; necrosis
Time Frame: 2 weeks
Population: 30 patients completed the 2 week timepoint of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Silverlon Arm
Number analyzed (Participants) | 30
Participants
  Grade 0 | 1
  Grade 1 | 20
  Grade 2 | 9
  Grade 3 | 0
  Grade 4 | 0

3. Secondary Outcome: Mean Radiation Induced Skin Reaction Assessment Scale
Description: This scoring system contains both a healthcare professions assessment scale and a patient symptom scale. The healthcare professional assessment scale (HPAS) individually scores the extent and severity of erythema, dry desquamation, moist desquamation, and necrosis using a 5-point scale from 0 to 4. Erythema is rated based on the degree of color change. Dry desquamation, moist desquamation, and necrosis are rated based on the percentage of the treatment area affected by that particular reaction. The HPAS score can range between 0 to 16. The patient symptom scale focuses on skin tenderness, itching, burning, and functional activity using a 4-point scale from 1 to 4. The patient symptom scale can range between 4 to 16. The Healthcare Professional Assessment Scale scores and the Patient Symptom Scale scores are added together for a total skin reaction score. The total skin reaction score can range between 4 to 32. The higher the score, the worse the skin reaction.
Time Frame: Mid study-visit, approximately 2 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Silverlon Arm
Number analyzed (Participants) | 30
score on a scale | 6.31 [5.47 to 6.94]

4. Secondary Outcome: Mean Radiation Induced Skin Reaction Assessment Scale
Description: This scoring system contains both a healthcare professions assessment scale and a patient symptom scale. The healthcare professional assessment scale (HAPS) individually scores the extent and severity of erythema, dry desquamation, moist desquamation, and necrosis using a 5-point scale from 0 to 4. Erythema is rated based on the degree of color change. Dry desquamation, moist desquamation, and necrosis are rated based on the percentage of the treatment area affected by that particular reaction. The HPAS score can range between 0 to 16. The patient symptom scale focuses on skin tenderness, itching, burning, and functional activity using a 4-point scale from 1 to 4. The patient symptom scale can range between 4 to 16. The Healthcare Professional Assessment Scale scores and the Patient Symptom Scale scores are added together for a total skin reaction score. The total skin reaction score can range between 4 to 32. The higher the score, the worse the skin reaction.
Time Frame: End of radiation therapy, approximately 4.5 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Silverlon Arm
Number analyzed (Participants) | 30
score on a scale | 10.77 [9.28 to 12.25]

5. Secondary Outcome: Mean Radiation Induced Skin Reaction Assessment Scale
Description: as for outcome 3
Time Frame: 2 weeks post radiation therapy, approximately 6.5 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Silverlon Arm
Number analyzed (Participants) | 30
score on a scale | 8.63 [7.39 to 9.87]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Silverlon Arm
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Silverlon Arm (N=31)
open area in inframammary fold (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT04238728/Prot_SAP_002.pdf
  • Informed Consent Form (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT04238728/ICF_001.pdf